CLINICAL TRIAL: NCT04471636
Title: Munich Remote SpO2 and Electrocardiogram Assessment in Covid-19 Patients
Brief Title: Telemedicine in Outpatient Covid-19 Patients
Acronym: COVID-SMART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Gesundheitsreferat (GSR), Landeshauptstadt München (Unknown); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Moritz F. Sinner, Assistant Professor, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-448
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Covid-19; Cardiovascular Risk Factor
Keywords: SARS-CoV2; Covid-19; cardiovascular disease; telemedicine; ECG; SpO2
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine Care (Experimental): Patients receive assessment at baseline and at 30 day follow up. Patient receive a smart watch capeable of recording SpO2, ECG, and heart rate. Patients also receive access to 24/7 medical hotline for telemedical care. All public services of the health care system remain available.
  Interventions: Device: Withings ScanWatch
- Control (No Intervention): Patients receive assessment at baseline and at 30 day follow up. Patient have access to all services of the health care system, but do not receive a smart watch or medical hotline access.

INTERVENTIONS:
Device: Withings ScanWatch — The smart watch is capable of recording SpO2, ECG, and heart rate.
  Arms: Telemedicine Care

SUMMARY:
Covid-19, a commonly severe respiratory tract infection caused by the SARS-CoV2 Coronavirus, poses an increasing threat to individual health and health care systems. The individual disease course ranges from mild to life threatening, the pandemic spread leads to a shortage of health care resources including intensive care availability. It should be the overarching goal to allocate sparse health care resources to those most at need and to simultaneously avoid unnecessary blocking of resources by clinically unjustified hospitalizations.

Individuals with preexisting cardiovascular conditions are at the highest risk of health deterioration, even at younger age. Objective criteria for hospitalization are not immediately available in a outpatient settings. Hence, hospitalization and emergency medical contact is often triggered by subjectively interpreted symptoms. The goal of this project is thus to improve the availability of objective measurements in the outpatient setting by means of an innovative, smartwatch mediated telemedicine approach.

To achieve this goal, the investigators will conduct a randomized clinical trial comparing a smartwatch based telemedicine intervention with standard of care. The intervention group will receive regular objective measurements of heart rate, ECG, and SpO2 and will get access to a 24/7 medical care hotline for consultation. The investigators hypothesize that the intervention group will benefit by a significant reduction in unnecessary hospitalizations and unplanned emergency medicine contacts.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV2 infection and clinical Covid-19 disease
* age ≥18 years
* Presence of ≥1 relevan cardiovascular condition, defined as (or):

  * atrial fibrillation
  * systolic or diastolic heart failure
  * LV ejection fraction <50%
  * coronary artery disease with past PCI or CABG
  * Past myocardial infarction
  * diabetes mellitus
  * arterial hypertension (treated or untreated)
  * active smoking
  * chronic obstructive lung disease
  * obesity (BMI ≥30kg/m2)
* availability of smartphone and sufficient internet connectivity at home
* ability to use smartwatch
* informed consent to study participation and data protection concept

Exclusion Criteria:

* Participation in concurrent clinical trial
* indication for hospitalization at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with a combination of hospitalization and unplanned use of hospital emergency department or emergency medical service | 30 days
  Occurrence of any of the above during follow-up

SECONDARY OUTCOMES:
Rate of participants hospitalized | 30 days
  Occurrence of hospitalization during follow-up
Rate of participants with unplanned use of hospital emergency department or emergency medical service | 30 days
  Occurrence of any of the above during follow-up
Rate of participants experiencing death of any cause | 30 days
  Occurrence of death of any cause during follow-up
Rate of participants experiencing death of Covid-19 | 30 days
  Occurence of daeth of Covid-19 during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Massberg, MD, Study Director — Department Head
Locations (1):
- LMU Klinikum, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Falkenhausen AS, Gail A, Geipel S, Scherer C, Stockhausen S, Sams LE, Becker F, Massberg S, Kaab S, Sinner MF. Symptoms of Depression and Anxiety After COVID-19 Despite Systematic Telemedical Care: Results From the Prospective COVID-SMART Study. Depress Anxiety. 2025 Apr 13;2025:9989990. doi: 10.1155/da/9989990. eCollection 2025. PMID 40259893